CLINICAL TRIAL: NCT03800641
Title: A Study of Dexmedetomidine Pharmacokinetics for Preoperative Sedation With Administration of Oral, Intravenous and Nasal Drops
Brief Title: A Study of Dexmedetomidine Pharmacokinetics for Preoperative Sedation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Jinhong Wu, Principal Investigator, Eye & ENT Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EyeEntFudan
Record Dates: First submitted 2019-01-07; First posted 2019-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Anxiety; Preoperative Care; Pharmacokinetics; Emergence Delirium
Keywords: Dexmedetomidine
MeSH Terms: conditions — Anxiety Disorders; Emergence Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- oral administration (Experimental): oral administration of dexmedetomidine 4μg/kg
  Interventions: Drug: Dexmedetomidine
- intravenous administration (Active Comparator): intravenous administration of dexmedetomidine 0.8μg/kg
  Interventions: Drug: Dexmedetomidine
- nasal administration (Experimental): nasal administration of dexmedetomidine 1μg/kg
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — oral, intravenous and nasal administration of Dexmedetomidine

SUMMARY:
Proper preoperative sedation can reduce patients' anxiety, enhance patients' cooperation and reduce perioperative complications. The investigators would explore the sedative effects of dexmedetomidine (DEX) with the administration of oral, intravenous and nasal drops, and detect DEX blood concentration in 15 participants, respectively. Pharmacokinetic parameters are detected at 8 time points ( before DEX administration, 10 min, 20 min, 30 min, 45 min, 60min, 90min and 120 min after administration). 3 ml arterial blood was collected at each time point. The blood samples are detected by mass spectrometer. The aim of this study is to investigate appropriate administration time and route for DEX sedation.

ELIGIBILITY:
Inclusion Criteria:

* 45 participants who undergo tympanoplasty would be enrolled after signment the informed consent.

Exclusion Criteria:

* The participants were excluded with any diseases about respiration, circulation, liver and kidney.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Dexmedetomidine pharmacokinetic curve | 120 min DEX pharmacokinetics
  Dexmedetomidine (DEX) blood concentration are detected at 8 time points (before DEX administration, 10 min, 20 min, 30 min, 45 min, 60min, 90min and 120 min after administration) in the groups of oral, intravenous and nasal drops administration of DEX. 3 ml arterial blood was collected at each time point. The blood samples are detected by mass spectrometer to detect blood concentration of DEX. Then DEX pharmacokinetic curve is made according to the DEX blood concentration.

SECONDARY OUTCOMES:
Effect of sedation | 10min after administration
  Evaluated with Ramsay sedation scale Score Response
  1. Anxious or restless or both
  2. Cooperative, orientated and tranquil
  3. Responding to commands
  4. Brisk response to stimulus
  5. Sluggish response to stimulus
  6. No response to stimulus
Evaluation of surgical field | 30min after administration
  Surgical field was evaluated according to the report Boezaart A.P.，van der Merwe J.，Coetzee A. Comparison of sodium nitroprusside- and esmolol-induced controlled hypotension for functional endoscopic sinus surgery. Can J Anaesth，1995，42(5 Pt 1): 373-376.
  0 No bleeding.
  1. Slight bleeding - no suctioning of blood required.
  2. Slight bleeding - occasional suctioning required. Surgical field not threatened.
  3. Slight bleeding - frequent suctioning required. Bleeding threatens surgical field a few seconds after suction is removed.
  4. Moderate bleeding - frequent suctioning required. Bleeding threatens surgical field directly after suction is removed.
  5. Severe bleeding - constant suctioning required. Bleeding appears faster than can be removed by suction. Surgical field severely threatened and surgery not possible.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye, Ear, Nose and Throat Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Wu J, Han Y, Lu Y, Zhuang Y, Li W, Jia J. Perioperative Low Dose Dexmedetomidine and Its Effect on the Visibility of the Surgical Field for Middle Ear Microsurgery: A Randomised Controlled Trial. Front Pharmacol. 2022 Feb 8;13:760916. doi: 10.3389/fphar.2022.760916. eCollection 2022. PMID 35211010